CLINICAL TRIAL: NCT06275776
Title: The Effect of Suturing Techniques on Aberrant Wound Recovery After Total Hip Arthroplasty
Brief Title: HIP-STITCH (Wound Recovery After THA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reinier Haga Orthopedisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OC-2022-005
Record Dates: First submitted 2024-02-05; First posted 2024-02-23 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Wound Healing Disturbance of
Keywords: Aberrant wound recovery; Total Hip Arthroplasty; Anterior approach; Monocryl Smooth Suture; Vicryl Rapide Braided Suture; Indermil Topical Skin Adhesive; Dermabond Prineo Skin Closure System; Stryker Zip Skin Closure System

STUDY DESIGN:
Intervention Model Description: Test subjects are randomised into one of four study arms. Each study arm corresponds with one of the suturing techniques that are going to be used to close the superficial skin after Total Hip Arthroplasty.
Who Masked: Outcomes Assessor
Masking Description: No one in this study can reasonably be blinded for the suturing technique during the duration of the study, since the suturing techniques differ substantially in shape, appearance and size. The only blinding in this study is the blinding of the outcome assessor to data of the test subjects. The assessor will only see the photographs of the wound/plaster, and the moment on which the photograph was taken. Additional information on the test subject, such as age, comorbidities, et cetera, will be withheld from the assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Monocryl Smooth Suture (Active Comparator): Study arm consisting of participants receiving Monocryl Smooth Suture for closure of the superficial skin. Monofilament suture, placed subcutaneously to approximate the wound edges. Currently used in standard care.
  Interventions: Device: Ethicon Monocryl Smooth Suture
- Vicryl Rapide + Indermil (Active Comparator): Study arm consisting of participants receiving Vicryl Rapide Braided Suture in combination with Indermil Topical Skin Adhesive for closure of the superficial skin. Multifilament suture, placed subcutaneously to approximate the wound edges. Skin glue is applied after the application of the suture to further seal the wound from the external environment. Currently used in standard care.
  Interventions: Device: Ethicon Vicryl Rapide Braided Suture; Device: Flexifuze Indermil Topical Skin Adhesive
- Dermabond Prineo (Experimental): Study arm consisting of participants receiving Dermabond Prineo Skin Closure System for closure of the superficial skin. Relatively novel skin closure system consisting of a self-adhesive transparent mesh, over which skin glue is applied as well. This system approximates the wound edges, shields the wound from the external environment, enables healthcare professionals to still be able to see the wound and surrounding tissue, and eliminates the invasive aspect of conventional sutures. Currently not used in standard care at the RHOC, but elsewhere it is being used.
  Interventions: Device: Dermabond Prineo Skin Closure System
- Stryker Zip (Experimental): Study arm consisting of participants receiving Stryker Zip Skin Closure System for closure of the superficial skin. Relatively novel skin closure system consisting of two self-adhesive strips placed parallel to either side of the wound. Zip tie/Cable tie-like structures running perpendicular to the adhesive strips can be tightened to approximate the wound edges and thusly close the wound. This system enables healthcare professionals to still see the wound and surrounding tissue, and eliminates the invasive aspect of conventional sutures. Currently not used in standard care at the RHOC, but elsewhere it is being used.
  Interventions: Device: Stryker Zip Skin Closure System

INTERVENTIONS:
Device: Ethicon Monocryl Smooth Suture — Monocryl Smooth Suture 3-0 antibacterial with PS-2 needle. Monofilament suture, placed subcutaneously to approximate the superficial wound edges. Currently used in standard care.
  Arms: Monocryl Smooth Suture
Device: Ethicon Vicryl Rapide Braided Suture — Vicryl Rapide Braided Suture 3-0 with FS-2 needle. Multifilament suture, placed subcutaneously to approximate the superficial wound edges. Currently used in standard care.
  Arms: Vicryl Rapide + Indermil
Device: Flexifuze Indermil Topical Skin Adhesive — Flexifuze Indermil Topical Skin Adhesive. The skin glue is applied after the application of the suture to further seal the wound from the external environment. Currently used in standard care.
  Arms: Vicryl Rapide + Indermil
Device: Dermabond Prineo Skin Closure System — Dermabond Prineo Skin Closure System. Novel skin closure system consisting of a self-adhesive transparent mesh, over which skin glue is applied as well. This system approximates the wound edges, shields the wound from the external environment, enables healthcare professionals to still see the wound and surrounding tissue, and eliminates the invasive aspect of conventional sutures. Currently not used in standard care at the RHOC, but elsewhere it is being used.
  Arms: Dermabond Prineo
Device: Stryker Zip Skin Closure System — Stryker Zip Skin Closure System. Novel skin closure system consisting of two self-adhesive strips placed parallel to either side of the wound. Zip tie/Cable tie-like structures running perpendicular to the adhesive strips can be tightened to approximate the wound edges and thusly close the wound. This system enables healthcare professionals to still see the wound and surrounding tissue, and eliminates the invasive aspect of conventional sutures. Currently not used in standard care at the RHOC, but elsewhere it is being used.
  Arms: Stryker Zip

SUMMARY:
This prospective randomised trial will investigate the effect of four different suturing techniques (Monocryl, Vicryl Rapide with Indermil skin glue, Dermabond Prineo, and Stryker Zip) on the amount of aberrant wound recovery within 14 days after total hip arthroplasty at the RHOC in Zoetermeer, The Netherlands.

This will be done by assessing photographs of the plaster and photographs of the operation wound with a self-developed classification model. The photographs of the plaster will be taken by the test subject at home at 3 days and 11 days postoperatively.

The photographs of the operation wound will be taken by a member of the research team, and the doctor's assistant, respectively, during a visit to the outpatient clinic at 7 days and 14 days postoperatively.

Hypothesis: Monocryl sutures give the highest amount of aberrant wound recovery within fourteen days after primary THA.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years or older.
* Scheduled to undergo Total Hip Arthroplasty via the anterior approach for any indication at the RHOC.
* No prior operations to the hip which is to be operated on.
* A good command of the Dutch language
* Able to give written informed consent.

Exclusion Criteria:

* Usage of cytostatics in the period ranging from fourteen days prior, to ninety days after the operation.
* Unable to, or difficulty with communicating in the Dutch language (e.g. due to mental disability, inability to understand/speak/write Dutch, et cetera).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Aberrant Wound Recovery | Up to fourteen days postoperatively
  Based on a self-developed classification model to assess the early wound recovery (within fourteen days postoperatively), a decision will be made whether the test subjects wound recovery is labelled as either ''normal wound recovery'', ''chance of aberrant wound recovery'', or ''aberrant wound recovery''.

SECONDARY OUTCOMES:
Number of Participants with Superficial or Deep Wound Infection | Up to ninety days postoperatively
  The amount of superficial or deep wound infections that occur in all the arms during the duration of the study. This will be assessed by checking the electronic patient file for contacts that might suggest infection, such as a DAIR, one-step exchange arthroplasty, two-step exchange arthroplasty, Girdlestone, or antibiotics usage. In addition to this, the questionnaire at fourteen days investigates whether the test subject has changed the adhesive plaster themselves at home. This is an indicator of wound fluid leakage, and thusly, might indicate infection.
Patient reported outcome measure: Satisfaction scores suturing method (Questionnaire) | Fourteen and ninety days postoperatively
  Questionnaire to be filled in by the participants. This self-developed questionnaire will assess the participants' satisfaction about the suturing method. This is not a standardised questionaire, as the investigators have developed it themselves.
  The satisfaction score will be assessed by means of two scale questions in the questionnaire. The first assessing patient reported satisfaction regarding the suturing technique ranging from one to ten (One being extremely dissatisfied, and ten being fully satisfied).
  The second question assesses how likely the participant is to recommend the suturing technique to a relative/friend/etc. from one to ten (One being highly unlikely, and ten being highly likely).
  A higher score on these questions corresponds with a higher satisfaction about the suturing technique. The participant has to pick one number on the scales corresponding to the satisfaction about the suturing technique, and the likelihood of recommendation.
Costs | Up to ninety days postoperatively.
  Total costs of the suturing method, including costs of the technique itself, time spend in the operating room, and also whether the test subject needs to visit the outpatient clinic visit for a control, or not.
  This will be done by assessing the costs of all these separate undertakings in standard care, and then adding the separate costs to the total costs. The theoretical costs will be enquired upon at the departments in the hospital which carry out these actions (i.e. outpatient clinic and operating room management), as well as the financial department of the hospital as a whole, who should be able to access this information.
Patient reported outcome measure: Score of Self-removal of the suturing technique (Questionnaire) | Fourteen days postoperatively
  This question will assess whether or not the test subject thinks he/she could have removed the suturing method himself/herself (or with aid of a friend/relative/etc.). This is not a standardised questionaire, as the investigators have developed it themselves.
  This is a scale question with possible answers ranging from one to ten, (One being extremely unlikely to remove the suturing technique, and ten being sure of removing it). A higher score on this question corresponds with a higher possibility of having removed the suturing technique themselves. The participant has to pick one number on the scale. The participant can also opt ''Not applicable in case he/she has received Monocryl (arm in the study). Clear instructions will be given in the questionnaire in order for the participant to know whether they have received this suturing technique or not.
  This is done to assess whether a patient would have to come to the outpatient clinic for a control appointment in standard care.
Patient reported outcome measure: Number of Participants with Other postoperative symptoms | Fourteen days and ninety days postoperatively
  Other symptoms which might have occurred postoperatively. These symptoms include fever, increase in pain, redness of the skin, pus coming from the wound, general feelings of discomfort, contact with the General Practitioner and antibiotics usage. This will be assessed by means of a questionnaire at fourteen en ninety days postoperatively.
Number and Type of Complications | Up to ninety days postoperatively
  Postoperative complications as recorded in the electronic patient file. Both the sheer number of complications will be registered per arm, as well as the type of complications that occur per arm.
Number of Visits to a Healthcare Professional | Up to ninety days postoperatively.
  Whether or not the participant has visited a healthcare professional postoperatively for wound-related causes. This number of times this occurs per arm will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan BW Vehmeijer, Dr., Principal Investigator — Reinier Haga Orthopedisch Centrum
Locations (1):
- Reinier Haga Orthopedisch Centrum, Zoetermeer, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No